CLINICAL TRIAL: NCT03920969
Title: Assessment of Self-esteem According to the Practice of a Sport Activity in a Population of Adults Living With HIV
Brief Title: Sport and Self Esteem in Patients Living With HIV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier le Mans (Other)
Collaborators: COordination REgionale de lutte contre les IST et le VIH (COREVIH) des Pays de la Loire (Unknown); Nantes University Hospital (Other); University Hospital, Angers (Other Government); Hospital, La Roche sur Yon (Unknown); Hospital, Saint Nazaire (Unknown); Centre Hospitalier de Cholet (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2018-S10/002
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: HIV Seropositivity
Keywords: Sport; HIV; Self Esteem
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Sports activity — Evaluation of physical activity using the International Physical Activity Questionnaire (IPAQ) short version.

SUMMARY:
Adapted athletic activity has shown benefits in patients with certain chronic diseases, including improving fatigue and pain in patients with cancer, and improving the symptoms of severe depression.

Among Patients Living with Human Immunodeficiency Virus (PLHIV), sport appears to be less common than for people who do not live with HIV. In fact, 44% of PLHIV in a Swiss cohort (10,500 patients) were inactive in 2014, whereas this percentage was 26% in the general population in Switzerland. We did not find any French data on the prevalence of sports activity among PLHIV.

The benefits of sport in PLHIV are numerous: meta-analyzes on interventional studies of aerobic and resistance exercises show a significant improvement in maximum oxygen consumption, muscle strength, percentage of body fat, quality of life and symptoms of depression. An improvement in cognitive function was noted in a randomized study. An Iranian randomized study of 2017 showed an improvement in the CD4 count, after 8 weeks of resistive exercise, but two meta-analyzes of 2016 and 2017 did not find a significant change in CD4 or viral load with physical exercise.

On the other hand, several studies have shown that sports practice improves self-esteem. In addition, an Australian randomized study in 2006 showed an improvement in self-efficacy in PLHIVs after a six-month exercise (aerobic and resistance) program. Furthermore, self-esteem (defined as positive self-esteem) is a factor facilitating adherence to antiretroviral therapy.

The objective of this descriptive study is to evaluate the prevalence of sports activity in a French adult population infected with HIV and to seek an association with self-esteem. In addition, the investigators will look for an association between sport and fatigue, pain, sleep, lymphocyte T CD4 cell levels, viral load.

ELIGIBILITY:
Inclusion Criteria:

* patient with HIV
* aged over 18
* Patient followed by a physician in one of the participating centers of the Regional coordination of the fight against HIV infection (COREVIH) Pays de la Loire

Exclusion Criteria:

* Refusal or unability to answer the self-questionnaire.
* Patient Under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all HIV-infected patients followed in one of the COREVIH centers of Pays de la Loire participating in this study. Participation in the study will be offered to patients during a usual visit as part of the follow-up of their pathology. The annual number of patients in 2017 being 4300, it is estimated that the number of patients included will be between 1000 and 2000 over 6 months of inclusion with a response rate of at least 50%.
Sampling Method: Non-Probability Sample
Enrollment: 1169 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of self-esteem according to the sport activity of PLHIV | six months
  Prevalence of self-esteem (Rosenberg questionnaire) among PLHIV, according to sport activity

SECONDARY OUTCOMES:
Description of the sporting activity of an adult HIV population | Six months
  Number and frequency of characteristics related to sports activity
Description of factors associated with sports activity: fatigue | Six months
  Prevalence of fatigue symptoms
Description of factors associated with sports activity: pain | Six months
  Prevalence of pain symptoms
Description of factors associated with sports activity: sleep | Six months
  Prevalence of sleep disorders
Search for a correlation between physical activity and HIV activity | 6 months
  Measure of the correlation between the measured physical activity and CD4 levels and HIV load.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Perez, MD, Principal Investigator — CH Le Mans
Locations (1):
- Centre Hospitalier Le Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: Undecided